CLINICAL TRIAL: NCT04075097
Title: Pain, Psychological, and Endocannabinoid Responses to Yoga in Breast Cancer Survivors With Chemotherapy-induced Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-1518; A176000 (Other: UW Madison); EDUC/KINESIOLOGY/KINESIOLOG (Other: UW Madison); UW18057 (Other: UWCCC)
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Neuropathic Pain
MeSH Terms: conditions — Breast Neoplasms; Neuralgia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The proposed study is an acute, single group, crossover pilot study where participants will complete two different experimental conditions: aerobic exercise and yoga.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): 44 minutes of moderate intensity walking on a treadmill.
  Interventions: Behavioral: Aerobic exercise
- Yoga (Experimental): 44 minutes of Iyengar yoga.
  Interventions: Behavioral: Iyengar yoga

INTERVENTIONS:
Behavioral: Aerobic exercise — 1 session
  Arms: Aerobic exercise
Behavioral: Iyengar yoga — 1 session
  Arms: Yoga

SUMMARY:
This study evaluates the acute effect of aerobic exercise and yoga on pain, plasma levels of endocannabinoids, and mood (i.e., mood disturbance and anxiety). Participants will complete three separate sessions on different days. The first session is a familiarization session in which participants complete questionnaires and are familiarized with the experimental protocols. During the second and third sessions, outcomes are measured before and after the participants complete either 44 minutes of moderate aerobic exercise (i.e., walking on a treadmill) or 44 minutes of yoga.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of breast cancer (stage 0-III),
* no evidence of active disease (i.e., recurrence, bone metastases, etc),
* presence of painful polyneuropathy, with onset coinciding or developing after receiving chemotherapy agents that in the opinion of the research team is likely to have caused such symptoms,
* at least six months since last active cancer treatment, with no further planned treatment (Note. active treatment is defined as surgery, chemotherapy, or radiation),
* the participant agrees to use the safety stop feature on the treadmill if needed,
* at least 18 years of age,
* and their physicians has provided consent for them to participate in yoga and aerobic exercise sessions.

Exclusion Criteria:

* Undergoing current chemotherapy or radiation treatment for cancer,
* taking anticoagulant therapy,
* uncontrolled medical conditions (i.e., uncontrolled hypertension, heart disease, stage 4 liver disease, end-stage renal disease, end-stage pulmonary disease, etc),
* stroke or myocardial infarction in the past 6 months,
* being pregnant or planning to become pregnant,
* severe mobility constraints (e.g., confined to a wheelchair),
* having a history of light headedness or fainting during blood draws or physical activity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Neuropathic Pain Sensations as determined by VAS | This will be measured 2 times during each experimental session- once before the assigned exercise task (i.e., baseline) and once upon task completion (i.e., approx. 50 mins later), approximately week 1 and week 2 on study.
  Visual analog scales (VAS) will be used to assess the intensity of the following sensations specific to neuropathic pain: pins and needles, tingles, stinging, and electrical pain sensations. The VAS is measured on a 100mm scale ranging from "No Pain" to "Worst Imaginable Pain."
Change in cold pain threshold | This will be measured 2 times during each experimental session- once before the assigned exercise task (i.e., baseline) and once upon task completion (i.e., approx. 50 mins later), approximately week 1 and week 2 on study.
  The minimum cold temperature needed to elicit a pain response.

SECONDARY OUTCOMES:
Change in total mood disturbance (Profile of Mood States) | This will be measured 2 times during each experimental session- once before the assigned exercise task (i.e., baseline) and once upon task completion (i.e., approx. 50 mins later), approximately week 1 and week 2 on study.
  65-item self-reported mood questionnaire that measures mood "right now." Scores range from 0-200 with higher scores indicating higher mood disturbance.
Change in plasma concentration of 2-Arachidonoylglycerol (2-AG) | This will be measured 2 times during each experimental session- once before the assigned exercise task (i.e., baseline) and once upon task completion (i.e., approx. 50 mins later), approximately week 1 and week 2 on study.
  Plasma concentration of 2-AG, one effector of the endocannabinoid system

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Koltyn, PhD, Principal Investigator — Professor of Kinesiology- Exercise Psychology, University of Wisconsin-Madison
Locations (1):
- University of Wisconsin-Madison Natatorium, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04075097/Prot_SAP_000.pdf